CLINICAL TRIAL: NCT00093262
Title: Efficacy Study of Clevidipine Assessing Its Postoperative Antihypertensive Effect in Cardiac Surgery (ESCAPE-2)
Brief Title: Study of Clevidipine Assessing Its Postoperative Antihypertensive Effect in Cardiac Surgery (ESCAPE-2)
Acronym: ESCAPE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMC-CLV-03-02; ESCAPE-2
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Postoperative Hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clevidipine (Experimental): Clevidipine was administered in a blinded fashion intravenously, starting with an infusion rate of 0.4 μg/kg/min (non weight-based equivalent is 2 mg/hr), titrating upward, as tolerated by the patient, in doubling increments approximately every 90 seconds up to an infusion rate of 3.2 μg/kg/min (16 mg/hr) to achieve the desired blood pressure-lowering effect. Up-titration to infusion rates above 3.2 μg/kg/min could be used, guided by the patient's response, by increasing the infusion rate in serial increments of 1.5 μg/kg/min, up to the maximum recommended clevidipine infusion rate of 8.0 μg/kg/min. Clevidipine was to be administered for a minimum of 30 minutes, unless bailout occurred, and up to a maximum of one hour.
  Interventions: Drug: clevidipine
- placebo (Placebo Comparator): Placebo consisted of 20% lipid emulsion (the same lipid vehicle used for clevidipine) administered in a blinded fashion intravenously following the same study drug administration guidelines as with clevidipine study drug administration guidelines. As with clevidipine, placebo was to be administered for a minimum of 30 minutes, unless bailout occurred, and up to a maximum of one hour.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clevidipine
  Other Names: clevidipine, Cleviprex
  Arms: clevidipine
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to establish the efficacy of of clevidipine versus placebo in treating postoperative hypertension. Approximately 100 patients with postoperative hypertension undergoing coronary artery bypass grafting (CABG), off-pump coronary artery bypass (OPCAB) or minimally invasive direct coronary artery bypass (MIDCAB) surgery and/or valve replacement/repair procedures were anticipated to be randomly assigned to one of two treatment groups: clevidipine or placebo.

DETAILED DESCRIPTION:
The primary objective was to determine the efficacy of clevidipine versus placebo in treating postoperative hypertension by comparing the incidence of bailout in the clevidipine and placebo treatment groups during the 30-minute time period from initiation of study drug. Secondary objectives included assessments of efficacy through measuring time to target blood pressure (BP) lowering effect defined as 15% reduction in SBP, change in mean arterial pressure (MAP) and the incidence of bailout by causality. Assessments for safety included change in heart rate (HR) from baseline.

ELIGIBILITY:
Pre-randomization Inclusion Criteria:

* Provide written informed consent before initiation of any study-related procedures.
* Be at least 18 years of age
* Be scheduled for cardiac surgery (including Coronary Artery Bypass Grafting [CABG], Off Pump Coronary Artery Bypass [OPCAB], Minimally Invasive Direct Coronary Artery Bypass [MIDCAB] surgery, and/or valve replacement/repair procedures)

Pre-randomization Exclusion Criteria:

* Women of child-bearing potential (unless they have a negative pregnancy test)
* Recent cerebrovascular accident (within 3 months before randomization)
* Known intolerance to calcium channel blockers
* Allergy to soybean oil or egg lecithin (components of the lipid vehicle)
* Pre-existing left bundle branch block or permanent ventricular pacing
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial.
* Participation in another therapeutic drug or therapeutic device trial within 30 days of starting study

Post-randomization Inclusion Criteria:

* Expected to survive beyond 24 hours post-surgical procedure
* No surgical complications or conditions, present or anticipated, that preclude them from inclusion in a double blind, placebo-controlled study
* Determined to be hypertensive (SBP > 140 mm Hg) within 4 hours of arrival in a postoperative setting
* It is the investigator's intent to lower the patient's SBP by a minimum of 15% from its baseline value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2003-12; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Incidence of bailout during 30-minute treatment period | During the first 30 minutes post study drug initiation
  The incidence of bailout defined as the premature and permanent discontinuation of study drug categorized according to the following reasons:
  * Bailout for lack of efficacy
  * Bailout for safety reason(s)
  * Bailout due to treatment failure

SECONDARY OUTCOMES:
Median time to target SBP lowering effect (defined as a reduction by 15% or more) | During the first 30 minutes post study drug initiation
Mean arterial pressure (MAP) change from baseline | During the first 30 minutes post study drug initiation
Heart rate change from baseline | During the first 30 minutes post study drug initiation
Incidence of bailout by causality | During the first 30 minutes post study drug initiation

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Discovery Alliance - Mobile Infirmary Medical Center, Mobile, Alabama
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - Stanford University School of Medicine, Stanford, California
  - Emory Hospital, Atlanta, Georgia
  - Heart Care Research Foundation, Blue Island, Illinois
  - MacNeal Hospital, Glencoe, Illinois
  - Wesley Medical Center, Wichita, Kansas
  - St. Lukes Hospital, Kansas City, Missouri
  - International Heart Institute, Missoula, Montana
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University - College of Physicians and Surgeons, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Discovery Alliance - Methodist Hospital / Diagnostic West Pavillion, Houston, Texas
  - Medical College of Wisconsin VAMC - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Singla N, Warltier DC, Gandhi SD, Lumb PD, Sladen RN, Aronson S, Newman MF, Corwin HL; ESCAPE-2 Study Group. Treatment of acute postoperative hypertension in cardiac surgery patients: an efficacy study of clevidipine assessing its postoperative antihypertensive effect in cardiac surgery-2 (ESCAPE-2), a randomized, double-blind, placebo-controlled trial. Anesth Analg. 2008 Jul;107(1):59-67. doi: 10.1213/ane.0b013e3181732e53. PMID 18635468